CLINICAL TRIAL: NCT03501953
Title: Neurophysiological Mechanisms of Physical Activity Interventions in Unique Environments
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not funded
Sponsor: Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NortheasternU
Record Dates: First submitted 2018-04-03; First posted 2018-04-18 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Environmental Exposure; Physical Activity
Keywords: Cognitive Change; Physical Activity; Environmental Exposure; Health Behavior
MeSH Terms: conditions — Motor Activity; Health Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two intervention classes that either take place outdoors or indoors. Intervention conditions are identical in protocol and measurements taken, and differ only in location of intervention.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature Exposure (Experimental): 6-week physical activity course in a natural environment
  Interventions: Behavioral: Physical Activity
- Urban Exposure (Active Comparator): 6-week physical activity course in an urban environment
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Six weeks of instructor-led physical activity sessions.

SUMMARY:
This randomized intervention is designed to compare the influence of physical activity in natural and urban environments on cognitive and physical health. Half of the participants will participate in a six-week physical activity class based in a natural environment, and half of the participants will participate in a six-week physical activity class based in an indoor environment. The investigators hypothesize the nature-based intervention will produce lower cognitive fatigue (measured using neurophysiological measurements), better cognitive performance (measured using cognitive assessments), and increased physical fitness (measuring using fitness testing).

DETAILED DESCRIPTION:
Research has yet to determine how regular physical activity in different environments influences physical and cognitive performance. Studies show exposure to natural environments can improve cognitive performance, increase creative thinking, and decrease stress-related responses. According to the theory of attention restoration, exposure to natural environments restores attentional resources because nature contains specific qualities that allow for directed attention to replenish and endorses health-related behaviors such as walking, running, and biking. Nature exposure is hypothesized to decrease activation of neural networks involved in cognitive control, therefore allowing for restoration of resources to occur. Activation of the cognitive control network is reflected through increased power of theta frequency (4-8 Hz) at the midfrontal regions (measured using electroencephalography; EEG), which reflects cognitive fatigue during rest. Previous research shows spending time in nature decreases midfrontal theta power, therefore reducing rumination and cognitive fatigue. Likewise, event-related potentials, such as higher P3 amplitude and shorter P3 latency during tasks, indicate better attentional allocation and processing speed, indicating better cognitive processing. These neurophysiological measurements are indicative of cognitive restoration and can determine changes in cognitive functioning over time.

The investigators propose to collect measurements of electroencephalography (spectral EEG, task-evoked event-related potentials), behavioral cognitive assessments (cognitive control, working memory performance), and health factors (VO2max) using a 2 (nature or urban physical activity intervention) x 2 (baseline and post-intervention sessions) design to determine changes in cognitive functioning across time. As part of an ongoing investigation in the cognitive and physical influence of intervention strategies, physical activity interventions will take place for a 6-week period, and participants will be recruited across three intervals of testing. Trained fitness instructors will lead participants in regularly scheduled 45-minute aerobic-based physical activity sessions three times a week. Each session will involve a combination of walking and running that progressively increases the duration of intensity throughout the 6-week period, starting at 20-minutes of moderate-to-vigorous training during the first week, and increasing duration by 5-minute intervals. Intervention groups will differ based on the location of the intervention. The nature-based intervention sessions will occur outdoors in a local public park in the Boston area. The urban-based intervention sessions will occur indoors in the Center for Cognitive & Brain Health intervention activity rooms.

ELIGIBILITY:
Inclusion Criteria:

* sedentary (1 or less exercise sessions per week)
* physically healthy
* normal or corrected-to-normal vision
* normal or corrected-to-normal hearing

Exclusion Criteria:

* currently treated for a neurological disorder
* currently treated for a physical health problem

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-15 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in spectral electroencephalography assessment at six weeks | six weeks from start of intervention
  Power at the midfrontal theta frequency
Changes from baseline in event-related potentials at six weeks | six weeks from start of intervention
  Stimulus-locked P3 component associated with the flanker task
Changes from baseline in cognitive assessment reaction time at six weeks | six weeks from start of intervention
  Reaction time on cognitive task
Changed from baseline in cardio-respiratory fitness assessment at six weeks | six weeks from start of intervention
  VO2max performance
Changes from baseline in cognitive assessment accuracy at six weeks | six weeks from start of intervention
  Accuracy score on cognitive task (0-100% score, higher accuracy is better)

SECONDARY OUTCOMES:
Accelerometry | 19 days
  number of steps and intensity of each session
Heart rate | 19 days
  average and max heart rate of each session

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hillman, Principal Investigator — Northeastern University; Arthur Kramer, Principal Investigator — Northeastern University

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- See also: Center for Cognitive and Brain Health — http://web.northeastern.edu/cbhlab/